CLINICAL TRIAL: NCT03846336
Title: An Investigation of Upper Extremity Function in Patients With Multiple Sclerosis, and Its Relation With Shoulder Position Sense and Disability Level
Brief Title: Upper Extremity Function, Shoulder Position Sense and Disability Level İn Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 25
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Physical Therapy; Upper Extremity Function; Position Sense
Keywords: Multiple Sclerosis; Upper Extremity Function; Position Sense
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Sclerosis (Experimental): Patients with confirmed diagnosis of clinically definite MS and physician-administered EDSS range of 1-3.5.
  Interventions: Other: Upper extremity function; Other: Shoulder position sense
- Healthy individuals (Other): 20 healthy volunteers with matching ages and genders.
  Interventions: Other: Upper extremity function; Other: Shoulder position sense

INTERVENTIONS:
Other: Upper extremity function — Upper extremity function was evaluated with 9-Hole Peg Test (9-HPT). The 9-HPT is a brief, standardized, quantitative test of upper extremity function. It consists of moving nine pegs into one of the nine holes on a peg board, then back into an open box. Both the dominant and non-dominant hands are tested twice.
Other: Shoulder position sense — Shoulder position sense was evaluated with a Dualer IQTM digital inclinometer (J-TECH medical, Salt Lake City, UT, USA). The absolute error scores (in degrees) for shoulder abduction and flexion at 30° and 60° was calculated. The upper extremity of the participant was positioned with the arm in the scapular plane for the abduction movement and in the sagittal plane for the flexion movement. After returning to the starting position, participants attempted to repeat the previously attained angle. Participants indicated verbally when they felt they had reached the angle and held their position. The measurement was repeated 2 more times for a total of 3 trials for each limb (non-dominant and dominant), with a 30-second rest period separating trials.

SUMMARY:
The purposes of this study is to investigate the relationship between upper extremity muscle function and shoulder position sense in patients with Multiple Sclerosis (MS) and which best projects the disability status.

Upper extremity dysfunction is considered to be the main cause of the loss performance of activities of daily living and this problem was include all motor and somatosensory components of function. Any failure in each of these components will likely create an impairment in the normal function.

One of the most important components of the somatosensory system is joint position sense, a sub-modality of proprioception. Position sense disorders are seen from the early stages of the disease and upper extremity function problems is experienced depending on position sense disorders in patients with MS.

Expanded Disability Status Scale (EDSS) is one of the most commonly outcome measures in evaluating the level of disability in MS population. Because EDSS scale emphasis on ambulation, so it is insensitive to upper extremity function. But the ability to use walking aids (e.g., canes, walkers, wheelchairs, etc.) may be affected by the UE impairment so shoulder position sense.

When literature is examined, there is no study which examines the relationship between upper extremity muscle function and shoulder position sense in patients with Multiple Sclerosis and which best projects the disability status. For all these reasons, we think that shoulder position sense is changed both dominant and non-dominant side during flexion and abduction movements in mild-moderate MS patients and that these deficits are correlated with upper extremity function and disability level.

DETAILED DESCRIPTION:
This study was aimed to investigate the relationship between upper extremity muscle function and shoulder position sense in patients with MS and which best projects the disability status.

21 PwMS and 20 healthy volunteers with matching ages and genders were included the study. A neurologic examination was performed using the EDSS by a neurologist.

Upper extremity function was evaluated with 9-Hole Peg Test (9-HPT). Shoulder position sense was evaluated with Dualer IQTM digital inclinometer (J-TECH medical, Salt Lake City, UK, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis Disease
* The level of disability should be between 0.5-4 according to EDSS

Exclusion Criteria:

* Patients with acute attacks (three months prior to the study)
* Mini-Mental State Examination (MMSE) score of less tahn 25 points
* History of shoulder injury, surgery, medical problems or other neurological disorders in any of the participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Upper extremity function | 1 month
  Upper extremity function was evaluated with the 9-Hole Peg Test (9-HPT). It consists of moving nine pegs into one of the nine holes on a peg board, then back into an open box. A stopwatch was used for the measurements and the scores were recorded in seconds (s).

SECONDARY OUTCOMES:
Shoulder position sense | 1 month
  Shoulder position sense was evaluated with a Dualer IQTM digital inclinometer (J-TECH medical, Salt Lake City, UT, USA).The absolute error scores (in degrees) for shoulder abduction and flexion at 30° and 60° was calculated. The difference between the target angle and the observed angle was calculated and the absolute error score was recorded by taking the average of 3 trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)

REFERENCES:
- [Derived] Unluer NO, Ozkan T, Yasa ME, Ates Y, Anlar O. An investigation of upper extremity function in patients with multiple sclerosis, and its relation with shoulder position sense and disability level. Somatosens Mot Res. 2019 Sep;36(3):189-194. doi: 10.1080/08990220.2019.1644998. Epub 2019 Aug 8. PMID 31393220